CLINICAL TRIAL: NCT01066819
Title: Prospective Observational Study on Predictors of Early On-treatment Response and Sustained Virological Response in a Cohort of Treatment naïve HCV-infected Patients Treated With Pegylated Interferons
Brief Title: PROPHESYS 3: Observational Study on Predictors of Response in Patients With Treatment-naïve Chronic Hepatitis C Initiated on Treatment With Pegasys (Peginterferon Alfa-2a) or Peginterferon-alfa-2b
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MV21542
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; peginterferon alfa-2b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort: Participants chronically infected with the hepatitis C virus including genotypes 1 to 6.
  Interventions: Drug: Peginterferon alfa-2a [Pegasys]; Drug: Peginterferon alfa-2b [PegIntron®]

INTERVENTIONS:
Drug: Peginterferon alfa-2a [Pegasys] — Peginterferon/ribavirin treatment period as prescribed by treating physician (e.g. 24 or 48 weeks) and treatment-free follow-up period of 24 weeks.
Drug: Peginterferon alfa-2b [PegIntron®] — Peginterferon/ribavirin treatment period as prescribed by treating physician (e.g. 24 or 48 weeks) and treatment-free follow-up period of 24 weeks.

SUMMARY:
This observational study will assess predictors of early on-treatment and sustained virological response in treatment-naïve patients with chronic hepatitis C initiated on treatment with Pegasys (peginterferon alfa-2a) or peginterferon alfa-2b and ribavirin. Data will be collected during the treatment period (24 or 48 weeks) and 12 and 24 weeks after the end of treatment. Target sample size is <2000.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/= 18 years of age
* chronic hepatitis C
* HIV HCV co-infection allowed
* informed consent to data collection

Exclusion Criteria:

* co-infection with Hepatitis B Virus (HBV)
* previous treatment with peginterferon and/or ribavirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving peginterferon alfa treatment at a medical centre
Sampling Method: Probability Sample
Enrollment: 1656 (Actual)
Dates: Start 2008-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (90):
- United States (89):
  - Birmingham, Alabama
  - Dothan, Alabama
  - Fresno, California
  - La Jolla, California
  - Lancaster, California
  - Loma Linda, California
  - Long Beach, California
  - Los Angeles, California
  - Sacramento, California
  - San Clemente, California
  - San Diego, California
  - San Francisco, California
  - San Mateo, California
  - Torrance, California
  - Aurora, Colorado
  - Hartford, Connecticut
  - Gainesville, Florida
  - Maitland, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Macon, Georgia
  - Marietta, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Opelousas, Louisiana
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Jackson, Mississippi
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Topeka, Missouri
  - Lebanon, New Hampshire
  - Egg Harbour Township, New Jersey
  - Hackensack, New Jersey
  - Hillsborough, New Jersey
  - Roseland, New Jersey
  - Voorhees Township, New Jersey
  - Albuquerque, New Mexico
  - Bayside, New York
  - Catskill, New York
  - Flushing, New York
  - New York, New York
  - Poughkeepsie, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Fayetteville, North Carolina
  - Rocky Mount, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Camp Hill, Pennsylvania
  - DuBois, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - West Nashville, Tennessee
  - Dallas, Texas
  - Galveston, Texas
  - Harlingen, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Huntington, West Virginia
  - Casper, Wyoming
- Santurce, Puerto Rico

REFERENCES:
- [Derived] Ferenci P, Aires R, Ancuta I, Arohnson A, Cheinquer H, Delic D, Gschwantler M, Larrey D, Tallarico L, Schmitz M, Tatsch F, Ouzan D. A tool for selecting patients with a high probability of sustained virological response to peginterferon alfa-2a (40kD)/ribavirin. Liver Int. 2014 Nov;34(10):1550-9. doi: 10.1111/liv.12439. Epub 2014 Jan 9. PMID 24329937

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1656 participants were enrolled in this study conducted from January 2008 to August 2011 at 111 centres in United States.
Groups:
- Genotype 1 (G1): Eligible participants with serologically proven Chronic hepatitis C (CHC) (Genotype 1) who received Pegylated Interferon (PEG-IFN) alfa-2a (PEGASYS®) or PEG-IFN alfa-2b (PegIntron®) plus ribavirin for up to 48 weeks according to the standard of care and in line with summaries of product characteristics (SPCs)/local labeling were observed.
- Genotype 2 (G2): Eligible participants with serologically proven CHC (Genotype 2) who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin for up to 48 weeks according to the standard of care and in line with SPCs/local labeling were observed.
- Genotype 3 (G3): Eligible participants with serologically proven CHC (Genotype 3) who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin for up to 48 weeks according to the standard of care and in line with SPCs/local labeling were observed.
- Genotype 4 (G4): Eligible participants with serologically proven CHC (Genotype 4) who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin for up to 48 weeks according to the standard of care and in line with SPCs/local labeling were observed.
- Genotype 5/6 (G5/6): Eligible participants with serologically proven CHC (Genotype 5/6) who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin for up to 48 weeks according to the standard of care and in line with SPCs/local labeling were observed.
- Genotype Unknown (UNK): Eligible participants with serologically proven CHC (Genotype unknown) who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin for up to 48 weeks according to the standard of care and in line with SPCs/local labeling were observed.
Period: Overall Study
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Started | 1006 | 348 | 257 | 25 | 7 | 13
Completed | 317 | 177 | 111 | 8 | 3 | 7
Not Completed | 689 | 171 | 146 | 17 | 4 | 6
Not completed — Adverse Event | 18 | 1 | 6 | 0 | 0 | 0
Not completed — Death | 5 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 22 | 1 | 2 | 1 | 0 | 0
Not completed — Physician Decision | 6 | 2 | 3 | 0 | 0 | 0
Not completed — Protocol Violation | 12 | 6 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 29 | 11 | 6 | 0 | 0 | 0
Not completed — Administrative | 6 | 4 | 2 | 0 | 0 | 0
Not completed — Not met inclusion/exclusion criteria | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Early termination | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Failed to return | 298 | 107 | 68 | 7 | 2 | 3
Not completed — Lab test not done | 9 | 0 | 2 | 1 | 0 | 0
Not completed — Miscellaneous | 28 | 10 | 18 | 1 | 0 | 0
Not completed — Non responders | 123 | 2 | 7 | 2 | 0 | 1
Not completed — Not categorised | 9 | 2 | 6 | 1 | 0 | 0
Not completed — Relapse | 16 | 4 | 3 | 0 | 0 | 0
Not completed — Results not available | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Screen failure | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Spontaneous cure | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Treatment never started | 85 | 19 | 19 | 3 | 2 | 2
Not completed — Treatment stopped | 12 | 1 | 2 | 1 | 0 | 0
Not completed — Other | 5 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The All Patient Enrolled Population included every participant of whom there was any data in the PROPHESYS database.
Groups:
- Genotype 1 (G1): Eligible participants with serologically proven CHC (Genotype 1) who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin for up to 48 weeks according to the standard of care and in line with SPCs/local labeling were observed.
- Total: Total of all reporting groups
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK) | Total
Number analyzed (Participants) | 1006 | 348 | 257 | 25 | 7 | 13 | 1656
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (9.68) | 49.7 (9.74) | 46.9 (9.41) | 46.4 (10.59) | 53.3 (10.48) | 45.6 (10.72) | 48.4 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 419 | 148 | 110 | 5 | 3 | 7 | 692
  Male | 587 | 200 | 147 | 20 | 4 | 6 | 964

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virological Response by Type of Peginterferon and Genotype in Modified All Treated Population
Description: Sustained virological response (SVR) was defined as virological response (VR) at 24 weeks after end of treatment (EOT). Virological response was defined as hepatitis C virus ribonucleic acid (HCV RNA) of <15 international units per milliliter (IU/mL) as assessed by COBAS AmpliPrep/COBAS TaqMan (CAP/CTM) or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (lower limit of detection [LLOD] 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The SVR is reported in treatment naive HCV mono-infected modified all-treated (mTRT) population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks (Wk) after EOT
Population: The mTRT population included all participants who received at least one dose of PEG-IFN and ribavirin, and had at least one post-baseline HCV RNA result. Participants with a baseline (BL) result <50 IU/mL were excluded. n = the number of participants analyzed at a given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Genotype 5/6 (G5/6): Participants with serologically proven CHC (Genotype 5/6) who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin for up to 48 weeks according to the standard of care and in line with SPCs/local labeling were observed.
- Genotype Unknown (UNK): Participants with serologically proven CHC (Genotype unknown) who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin for up to 48 weeks according to the standard of care and in line with SPCs/local labeling were observed.
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 674 | 267 | 188 | 18 | 3 | 2
percentage of participants
  Peg IFN Alfa 2a (n=568,221,159,16,2,1) | 30.3 [26.5 to 34.2] | 55.7 [48.8 to 62.3] | 43.4 [35.6 to 51.5] | 31.3 [11.0 to 58.7] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 97.5]
  Peg IFN Alfa 2b (n=106,46,29,2,1,1) | 23.6 [15.9 to 32.8] | 50.0 [34.9 to 65.1] | 37.9 [20.7 to 57.7] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 97.5]

2. Primary Outcome: Percentage of Participants With Sustained Virological Response by Type of Peginterferon and Genotype in Per Protocol Population
Description: Sustained virological response was defined as VR at 24 weeks after EOT. Virological response was defined as HCV RNA of <15 IU/mL as assessed by CAP/CTM or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (LLOD 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The SVR is reported in treatment naive HCV mono-infected per protocol (PP) population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: The per-protocol (PP) population included all participants who met the inclusion and exclusion criteria of the study. n = the number of participants analyzed at a given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 564 | 231 | 151 | 16 | 3 | 2
percentage of participants
  Peg IFN Alfa 2a (n=476,190,123,14,2,1) | 31.5 [27.4 to 35.9] | 57.4 [50.0 to 64.5] | 48.8 [39.7 to 58.0] | 35.7 [12.8 to 64.9] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 97.5]
  Peg IFN Alfa 2b (n=88,41,28,2,1,1) | 26.1 [17.3 to 36.6] | 48.8 [32.9 to 64.9] | 35.7 [18.6 to 55.9] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 97.5]

3. Primary Outcome: Percentage of Participants With Modified Sustained Virological Response Over Time by Type of Peginterferon and Genotype in Modified All Treated Population
Description: Modified sustained virological response (mSVR) was defined as modified virological response (mVR) of HCV RNA <50 IU/mL at 24 weeks after EOT. The mSVR is reported in treatment naive HCV mono-infected mTRT population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: The mTRT population included all participants who received at least one dose of PEG-IFN and ribavirin, and had at least one post-baseline HCV RNA result. Participants with a baseline result <50 international units per millilitre (IU/mL) were excluded. n = the number of participants analyzed at a given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 674 | 267 | 188 | 18 | 3 | 2
percentage of participants
  Peg IFN Alfa 2a (n=568,221,159,16,2,1) | 30.6 [26.9 to 34.6] | 56.1 [49.3 to 62.8] | 43.4 [35.6 to 51.5] | 31.3 [11.0 to 58.7] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 97.5]
  Peg IFN Alfa 2b (n=106,46,29, 2,1,1) | 23.6 [15.9 to 32.8] | 50.0 [34.9 to 65.1] | 37.9 [20.7 to 57.7] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 97.5]
Statistical Analysis 1: Comparison: Genotype 1 (G1); The statistical analysis is presented for Ethnic origin (ASIAN vs WHITE/CAUCASIAN). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week [Wk] 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0045, Regression, Logistic; Odds Ratio (OR) = 5.596, 95% CI 2-sided [1.704 to 18.378]
Statistical Analysis 2: Comparison: Genotype 1 (G1); The statistical analysis is presented for Ethnic origin (BLACK vs WHITE/CAUCASIAN). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.9755, Regression, Logistic; Odds Ratio (OR) = 0.989, 95% CI 2-sided [0.497 to 1.967]
Statistical Analysis 3: Comparison: Genotype 1 (G1); The statistical analysis is presented for Ethnic origin (HISPANIC vs WHITE/CAUCASIAN). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.4786, Regression, Logistic; Odds Ratio (OR) = 0.743, 95% CI 2-sided [0.327 to 1.688]
Statistical Analysis 4: Comparison: Genotype 1 (G1); The statistical analysis is presented for Ethnic origin (OTHER vs WHITE/CAUCASIAN). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0140, Regression, Logistic; Odds Ratio (OR) = 5.380, 95% CI 2-sided [1.405 to 20.597]
Statistical Analysis 5: Comparison: Genotype 1 (G1); The statistical analysis is presented for treatment duration after VR in weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.078, 95% CI 2-sided [1.062 to 1.094]
Statistical Analysis 6: Comparison: Genotype 1 (G1); The statistical analysis is presented for Ethnic origin (ASIAN vs WHITE/CAUCASIAN). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0035, Regression, Logistic; Odds Ratio (OR) = 6.136, 95% CI 2-sided [1.819 to 20.701]
Statistical Analysis 7: Comparison: Genotype 1 (G1); The statistical analysis is presented for Ethnic origin (BLACK vs WHITE/CAUCASIAN). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.7821, Regression, Logistic; Odds Ratio (OR) = 0.903, 95% CI 2-sided [0.439 to 1.857]
Statistical Analysis 8: Comparison: Genotype 1 (G1); The statistical analysis is presented for Ethnic origin (HISPANIC vs WHITE/CAUCASIAN). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.4846, Regression, Logistic; Odds Ratio (OR) = 0.740, 95% CI 2-sided [0.317 to 1.723]
Statistical Analysis 9: Comparison: Genotype 1 (G1); The statistical analysis is presented for Ethnic origin (OTHER vs WHITE/CAUCASIAN). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0170, Regression, Logistic; Odds Ratio (OR) = 5.424, 95% CI 2-sided [1.353 to 21.749]
Statistical Analysis 10: Comparison: Genotype 1 (G1); The statistical analysis is presented for HCV RNA at BL in log10(IU/mL). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0125, Regression, Logistic; Odds Ratio (OR) = 0.695, 95% CI 2-sided [0.523 to 0.925]
Statistical Analysis 11: Comparison: Genotype 1 (G1); The statistical analysis is presented for average number of drinks per week (1 vs 0). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0139, Regression, Logistic; Odds Ratio (OR) = 3.472, 95% CI 2-sided [1.288 to 9.357]
Statistical Analysis 12: Comparison: Genotype 1 (G1); The statistical analysis is presented for average number of drinks per week (> 1 vs 0). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.6327, Regression, Logistic; Odds Ratio (OR) = 1.179, 95% CI 2-sided [0.601 to 2.311]
Statistical Analysis 13: Comparison: Genotype 1 (G1); The statistical analysis is presented for treatment duration after VR in weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.061, 95% CI 2-sided [1.042 to 1.080]
Statistical Analysis 14: Comparison: Genotype 1 (G1); The statistical analysis is presented for Cumulative PEG-IFN alfa-2a dose per 1000 ug. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0033, Regression, Logistic; Odds Ratio (OR) = 1.185, 95% CI 2-sided [1.058 to 1.326]
Statistical Analysis 15: Comparison: Genotype 2 (G2); [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.227, 95% CI 2-sided [1.151 to 1.308]
Statistical Analysis 16: Comparison: Genotype 2 (G2); The statistical analysis is presented for cumulative ribavirin dose per 10000 mg, 1st 12 weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0289, Regression, Logistic; Odds Ratio (OR) = 0.814, 95% CI 2-sided [0.676 to 0.979]
Statistical Analysis 17: Comparison: Genotype 2 (G2); [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.276, 95% CI 2-sided [1.177 to 1.383]
Statistical Analysis 18: Comparison: Genotype 2 (G2); The statistical analysis is presented for Cumulative ribavirin dose per 10000 mg. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0099, Regression, Logistic; Odds Ratio (OR) = 0.894, 95% CI 2-sided [0.821 to 0.973]
Statistical Analysis 19: Comparison: Genotype 3 (G3); The statistical analysis is presented for age per 10 years. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0058, Regression, Logistic; Odds Ratio (OR) = 1.945, 95% CI 2-sided [1.213 to 3.120]
Statistical Analysis 20: Comparison: Genotype 3 (G3); [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.262, 95% CI 2-sided [1.154 to 1.380]
Statistical Analysis 21: Comparison: Genotype 3 (G3); The statistical analysis is presented for age per 10 years. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0058, Regression, Logistic; Odds Ratio (OR) = 1.945, 95% CI 2-sided [1.213 to 3.120]
Statistical Analysis 22: Comparison: Genotype 3 (G3); [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.262, 95% CI 2-sided [1.154 to 1.380]
Statistical Analysis 23: Comparison: Genotype 1 (G1); The statistical analysis is presented for Ethnic origin (ASIAN vs WHITE/CAUCASIAN). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0205, Regression, Logistic; Odds Ratio (OR) = 3.615, 95% CI 2-sided [1.219 to 10.721]
Statistical Analysis 24: Comparison: Genotype 1 (G1); The statistical analysis is presented for Ethnic origin (BLACK vs WHITE/CAUCASIAN). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.9557, Regression, Logistic; Odds Ratio (OR) = 0.981, 95% CI 2-sided [0.506 to 1.903]
Statistical Analysis 25: Comparison: Genotype 1 (G1); The statistical analysis is presented for Ethnic origin (HISPANIC vs WHITE/CAUCASIAN). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.2000, Regression, Logistic; Odds Ratio (OR) = 0.599, 95% CI 2-sided [0.273 to 1.312]
Statistical Analysis 26: Comparison: Genotype 1 (G1); The statistical analysis is presented for (OTHER vs WHITE/CAUCASIAN). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0437, Regression, Logistic; Odds Ratio (OR) = 3.684, 95% CI 2-sided [1.037 to 13.083]
Statistical Analysis 27: Comparison: Genotype 1 (G1); The statistical analysis is presented for On-treatment response (RVR vs NO RVR/EVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 134.60, 95% CI 2-sided [17.956 to 1009.0]
Statistical Analysis 28: Comparison: Genotype 1 (G1); The statistical analysis is presented for On-treatment response (cEVR vs NO RVR/EVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 77.905, 95% CI 2-sided [10.521 to 576.85]
Statistical Analysis 29: Comparison: Genotype 1 (G1); The statistical analysis is presented for On-treatment response (pEVR vs NO RVR/EVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0105, Regression, Logistic; Odds Ratio (OR) = 14.527, 95% CI 2-sided [1.872 to 112.73]
Statistical Analysis 30: Comparison: Genotype 2 (G2); The statistical analysis is presented for age per 10 years. The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0041, Regression, Logistic; Odds Ratio (OR) = 1.563, 95% CI 2-sided [1.152 to 2.120]
Statistical Analysis 31: Comparison: Genotype 2 (G2); The statistical analysis is presented for On-treatment response, combined (RVR vs NO RVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 5.557, 95% CI 2-sided [2.405 to 12.838]
Statistical Analysis 32: Comparison: Genotype 3 (G3); [analysis description as in outcome 3, analysis 30]; Test type: Superiority or Other; p = 0.0037, Regression, Logistic; Odds Ratio (OR) = 1.822, 95% CI 2-sided [1.216 to 2.732]
Statistical Analysis 33: Comparison: Genotype 3 (G3); [analysis description as in outcome 3, analysis 31]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 11.342, 95% CI 2-sided [3.977 to 32.347]
Statistical Analysis 34: Comparison: Genotype 1 (G1); The statistical analysis is presented for treatment duration after VR in weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2b; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.112, 95% CI 2-sided [1.068 to 1.158]
Statistical Analysis 35: Comparison: Genotype 1 (G1); The statistical analysis is presented for treatment duration after VR in weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2b; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.112, 95% CI 2-sided [1.068 to 1.158]
Statistical Analysis 36: Comparison: Genotype 1 (G1); The statistical analysis is presented for On-treatment response, combined (RVR vs NO RVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2b; Test type: Superiority or Other; p = 0.0035, Regression, Logistic; Odds Ratio (OR) = 4.921, 95% CI 2-sided [1.686 to 14.362]

4. Primary Outcome: Percentage of Participants With Modified Sustained Virological Response by Type of Peginterferon and Genotype in Per Protocol Population
Description: Modified sustained virological response is defined as mVR of HCV RNA <50 IU/mL at 24 weeks after EOT. The mSVR is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: The PP population included all participants who met the inclusion and exclusion criteria of the study. n = the number of participants analyzed at a given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 564 | 231 | 151 | 16 | 3 | 2
percentage of participants
  Peg IFN Alfa 2a (n=476,190,123,14,2,1) | 31.9 [27.8 to 36.3] | 57.9 [50.5 to 65.0] | 48.8 [39.7 to 58.0] | 35.7 [12.8 to 64.9] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 97.5]
  Peg IFN Alfa 2b (n=88,41,28,2,1,1) | 26.1 [17.3 to 36.6] | 48.8 [32.9 to 64.9] | 35.7 [18.6 to 55.9] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 97.5]

5. Primary Outcome: Percentage of Participants With Predictive Values of Virological Response by Week 4 and 12 on Modified Sustained Virological Response After Treatment Initiation in Modified All Treated Population
Description: The probability that a participant who developed VR by Week 4 and 12 and also achieved mSVR at 24 weeks after EOT was called the positive predictive value (PPV) of the VR by Wk 4 for mSVR. The probability that a participant who failed to develop VR by Wk 4 and 12 and also failed to achieve mSVR at 24 weeks after EOT was called the negative predictive value (NPV) of the VR by Wk 4 and 12 for mSVR. Predictive values of VR are reported in treatment naive HCV mono-infected mTRT participants who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: The mTRT population included all participants who received at least one dose of PEG-IFN and ribavirin, and had at least one post-baseline HCV RNA result. Participants with a baseline result <50 IU/mL were excluded. n = the number of participants analyzed at a given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 674 | 267 | 188 | 18 | 3 | 2
percentage of participants
  Wk4,PegIFNAlfa2a,PPV (n=568,221,159,16,2,1) | 53.8 [44.9 to 62.6] | 62.0 [54.5 to 69.0] | 56.1 [46.5 to 65.4] | 20.0 [0.5 to 71.6] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk4, PegIFNAlfa2a,NPV (n=568,221,159,16,2,1) | 76.7 [72.3 to 80.7] | 78.1 [60.0 to 90.7] | 88.1 [74.4 to 96.0] | 60.0 [26.2 to 87.8] | 0.0 [0.0 to 97.5] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk4, PegIFNAlfa2b, PPV (n=106,46,29,2,1,1) | 52.6 [28.9 to 75.6] | 52.6 [35.8 to 69.0] | 50.0 [27.2 to 72.8] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk4, PegIFNAlfa2b, NPV (n=106,46,29,2,1,1) | 81.6 [71.0 to 89.5] | 57.1 [18.4 to 90.1] | 87.5 [47.3 to 99.7] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk12,PegIFNAlfa2a,PPV (n=568,221,159,16,2,1) | 48.4 [42.7 to 54.1] | 59.0 [52.1 to 65.8] | 51.1 [42.3 to 59.9] | 50.0 [18.7 to 81.3] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 97.5]
  Wk12,PegIFNAlfa2a, NPV(n=568,221,159,16,2,1) | 91.3 [87.1 to 94.5] | 100.0 [71.5 to 100.0] | 95.8 [78.9 to 99.9] | 100.0 [47.8 to 100.0] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk12,PegIFNAlfa2b, PPV (n=106,46,29,2,1,1) | 52.4 [36.4 to 68.0] | 50.0 [34.6 to 65.4] | 40.7 [22.4 to 61.2] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk12, PegIFNAlfa2b, NPV (n=106, 46,29, 2,1,1) | 96.6 [88.3 to 99.6] | 50.0 [1.3 to 98.7] | 100.0 [15.8 to 100.0] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.

6. Primary Outcome: Percentage of Participants With Predictive Values of Virological Response by Week 4 and 12 on Modified Sustained Virological Response After Treatment Initiation in Per Protocol Population
Description: The probability that a participant who developed VR by Week 4 and 12 and also achieved mSVR at 24 weeks after EOT was called the PPV of the VR by Wk 4 for mSVR. The probability that a participant who failed to develop VR by Wk 4 and 12 and also failed to achieve mSVR at 24 weeks after EOT was called the NPV of the VR by Wk 4 and 12 for mSVR. Predictive values of VR are reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 564 | 231 | 151 | 16 | 3 | 2
percentage of participants
  Wk4,PegIFNAlfa2a,PPV (n=476,190,123,14,2,1) | 54.1 [44.3 to 63.7] | 62.4 [54.6 to 69.8] | 55.0 [44.7 to 65.0] | 20.0 [0.5 to 71.6] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk4, PegIFNAlfa2a,NPV (n=476,190,123,14,2,1) | 75.4 [70.5 to 79.8] | 70.8 [48.9 to 87.4] | 77.3 [54.6 to 92.2] | 50.0 [15.7 to 84.3] | 0.0 [0.0 to 97.5] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk4, PegIFNAlfa2b, PPV (n=88,41,28,2,1,1) | 50.0 [24.7 to 75.3] | 51.5 [33.5 to 69.2] | 47.4 [24.4 to 71.1] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk4, PegIFNAlfa2b, NPV (n=88,41,28,2,1,1) | 78.1 [66.0 to 87.5] | 57.1 [18.4 to 90.1] | 87.5 [47.3 to 99.7] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk12,PegIFNAlfa2a,PPV (n=476,190,123,14,2,1) | 49.6 [43.4 to 55.8] | 59.1 [51.7 to 66.3] | 51.3 [41.8 to 60.7] | 50.0 [18.7 to 81.3] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 97.5]
  Wk12,PegIFNAlfa2a, NPV(n=476, 190,123,14,2,1) | 90.5 [85.7 to 94.1] | 100.0 [39.8 to 100.0] | 87.5 [47.3 to 99.7] | 100.0 [29.2 to 100.0] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk12,PegIFNAlfa2b, PPV (n=88,41,28,2,1,1) | 55.6 [38.1 to 72.1] | 48.7 [32.4 to 65.2] | 38.5 [20.2 to 59.4] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk12, PegIFNAlfa2b, NPV (n=88,41,28,2,1,1) | 95.8 [85.7 to 99.5] | 50.0 [1.3 to 98.7] | 100.0 [15.8 to 100.0] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.

7. Secondary Outcome: Percentage of Participants With Virological Response by Type of Peginterferon and Genotype in Modified All Treated Population Over Time
Description: Virological Response (VR) was defined as HCV RNA <15 IU/mL as assessed by COBAS AmpliPrep/COBAS TaqMan (HCV) (CAP/CTM) or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (lower limit of detection 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. PEOT= Post End of Treatment. EOT= 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At Week 2, Week 4, Week 12, EOT, and at 12 Weeks after EOT
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 674 | 267 | 188 | 18 | 3 | 2
percentage of participants
  Wk2,PegIFNAlfa2a (n=568,221,159 ,16,2,1) | 6.5 [4.6 to 8.9] | 25.8 [20.2 to 32.1] | 20.8 [14.7 to 27.9] | 12.5 [1.6 to 38.3] | 0.0 [0.0 to 84.2] | 100.0 [2.5 to 100.0]
  Wk2,PegIFNAlfa2b (n=106,46,29,2,1,1) | 2.8 [0.6 to 8.0] | 17.4 [7.8 to 31.4] | 24.1 [10.3 to 43.5] | 0.0 [0.0 to 84.2] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk4,PegIFNAlfa2a (n=568,221,159,16,2,1) | 22.9 [19.5 to 26.6] | 83.3 [77.7 to 87.9] | 71.7 [64.0 to 78.5] | 31.3 [11.0 to 58.7] | 50.0 [1.3 to 98.7] | 100.0 [2.5 to 100.0]
  Wk4,PegIFNAlfa2b (n=106,46,29,2,1,1) | 17.9 [11.2 to 26.6] | 82.6 [68.6 to 92.2] | 69.0 [49.2 to 84.7] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk12,PegIFNAlfa2a (n=568,221,159,16,2,1) | 54.9 [50.7 to 59.1] | 95.0 [91.3 to 97.5] | 83.6 [77.0 to 89.0] | 62.5 [35.4 to 84.8] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk12,PegIFNAlfa2b (n=106,46,29,2,1,1) | 39.6 [30.3 to 49.6] | 95.7 [85.2 to 99.5] | 93.1 [77.2 to 99.2] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  EOT,PegIFNAlfa2a (n=568,221,159,16,2,1) | 55.3 [51.1 to 59.4] | 85.5 [80.2 to 89.9] | 74.2 [66.7 to 80.8] | 56.3 [29.9 to 80.2] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  EOT,PegIFNAlfa2b (n=106,46,29,2,1,1) | 38.7 [29.4 to 48.6] | 84.8 [71.1 to 93.7] | 72.4 [52.8 to 87.3] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  12Wk PEOT,PegIFNAlfa2a (n=568,221,159,16,2,1) | 34.5 [30.6 to 38.6] | 59.7 [52.9 to 66.3] | 48.4 [40.4 to 56.5] | 31.3 [11.0 to 58.7] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  12Wk PEOT,PegIFNAlfa2b (n=106,46,29,2,1,1) | 29.2 [20.8 to 38.9] | 54.3 [39.0 to 69.1] | 44.8 [26.4 to 64.3] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 97.5]

8. Secondary Outcome: Percentage of Participants With Virological Response by Type of Peginterferon and Genotype in Per Protocol Population Over Time
Description: Virological response (VR) was defined as HCV RNA <15 IU/mL as assessed by CAP/CTM or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (LLOD 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The VR is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment. PEOT= Post End of Treatment
Time Frame: At Week 2, Week 4, Week 12, EOT, and at 12 Weeks after EOT
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 564 | 231 | 151 | 16 | 3 | 2
percentage of participants
  Wk2,PegIFNAlfa2a (n=476,190,123,14,2,1) | 7.4 [5.2 to 10.1] | 28.9 [22.6 to 36.0] | 23.6 [16.4 to 32.1] | 14.3 [1.8 to 42.8] | 0.0 [0.0 to 84.2] | 100.0 [2.5 to 100.0]
  Wk2,PegIFNAlfa2b (n=88,41,28,2,1,1) | 3.4 [0.7 to 9.6] | 19.5 [8.8 to 34.9] | 25.0 [10.7 to 44.9] | 0.0 [0.0 to 84.2] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk4,PegIFNAlfa2a (n=476,190,123,14,2,1) | 22.9 [19.2 to 26.9] | 86.8 [81.2 to 91.3] | 81.3 [73.3 to 87.8] | 35.7 [12.8 to 64.9] | 50.0 [1.3 to 98.7] | 100.0 [2.5 to 100.0]
  Wk4,PegIFNAlfa2b (n=88,41,28,2,1,1) | 18.2 [10.8 to 27.8] | 80.5 [65.1 to 91.2] | 67.9 [47.6 to 84.1] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk12,PegIFNAlfa2a (n=476,190,123,14,2,1) | 55.5 [50.9 to 60.0] | 97.9 [94.7 to 99.4] | 93.5 [87.6 to 97.2] | 71.4 [41.9 to 91.6] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk12,PegIFNAlfa2b (n=88,41,28,2,1,1) | 40.9 [30.5 to 51.9] | 95.1 [83.5 to 99.4] | 92.9 [76.5 to 99.1] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  EOT,PegIFNAlfa2a (n=476,190,123,14,2,1) | 55.5 [50.9 to 60.0] | 88.9 [83.6 to 93.0] | 81.3 [73.3 to 87.8] | 64.3 [35.1 to 87.2] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  EOT,PegIFNAlfa2b (n=88,41,28,2,1,1) | 43.2 [32.7 to 54.2] | 85.4 [70.8 to 94.4] | 71.4 [51.3 to 86.8] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk12 PEOT,PegIFNAlfa2a (n=476,190,123,14,2,1) | 35.5 [31.2 to 40.0] | 62.1 [54.8 to 69.0] | 52.8 [43.6 to 61.9] | 35.7 [12.8 to 64.9] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk12 EOT,PegIFNAlfa2b (n=88,41,28,2,1,1) | 30.7 [21.3 to 41.4] | 51.2 [35.1 to 67.1] | 42.9 [24.5 to 62.8] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]

9. Secondary Outcome: Percentage of Participants With Modified Virological Response by Type of Peginterferon and Genotype in Modified All Treated Population Over Time
Description: Modified virological response (mVR) was defined as HCV RNA <50 IU/mL as assessed by CAP/CTM or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (LLOD 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The mVR is reported in treatment naive HCV mono-infected mTRT population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment. PEOT= Post End of Treatment
Time Frame: At Week 2, Week 4, Week 12, EOT, and at 12 Weeks after EOT
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 674 | 267 | 188 | 18 | 3 | 2
percentage of participants
  Wk2, Peg IFN Alfa 2a (n=568,221,159,16,2,1) | 7.6 [5.5 to 10.1] | 28.5 [22.7 to 34.9] | 25.8 [19.2 to 33.3] | 18.8 [4.0 to 45.6] | 50.0 [1.3 to 98.7] | 100.0 [2.5 to 100.0]
  Wk2, Peg IFN Alfa 2b (n=106,46,29,2,1,1) | 3.8 [1.0 to 9.4] | 19.6 [9.4 to 33.9] | 31.0 [15.3 to 50.8] | 0.0 [0.0 to 84.2] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk4, Peg IFN Alfa 2a (n=568,221,159,16,2,1) | 25.9 [22.3 to 29.7] | 85.5 [80.2 to 89.9] | 75.5 [68.0 to 81.9] | 37.5 [15.2 to 64.6] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk4, Peg IFN Alfa 2b (n=106,46,29,2,1,1) | 22.6 [15.1 to 31.8] | 84.8 [71.1 to 93.7] | 75.9 [56.5 to 89.7] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk12, Peg IFN Alfa 2a (n=568,221,159,16,2,1) | 58.1 [53.9 to 62.2] | 95.5 [91.8 to 97.8] | 85.5 [79.1 to 90.6] | 62.5 [35.4 to 84.8] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk12,Peg IFN Alfa 2b (n=106,46,29,2,1,1) | 43.4 [33.8 to 53.4] | 95.7 [85.2 to 99.5] | 93.1 [77.2 to 99.2] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  EOT, Peg IFN Alfa 2a (n=568,221,159,16,2,1) | 56.2 [52.0 to 60.3] | 86.9 [81.7 to 91.0] | 75.5 [68.0 to 81.9] | 56.3 [29.9 to 80.2] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  EOT, Peg IFN Alfa 2b (n=106,46,29,2,1,1) | 40.6 [31.1 to 50.5] | 87.0 [73.7 to 95.1] | 72.4 [52.8 to 87.3] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  12wk PEOT,PegIFNAlfa2a(n=568,221,159,16,2,1) | 34.9 [30.9 to 38.9] | 60.6 [53.9 to 67.1] | 48.4 [40.4 to 56.5] | 37.5 [15.2 to 64.6] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  12wk PEOT, PegIFNAlfa2b(n=106,46,29,2,1,1) | 29.2 [20.8 to 38.9] | 54.3 [39.0 to 69.1] | 44.8 [26.4 to 64.3] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 97.5]

10. Secondary Outcome: Percentage of Participants With Modified Virological Response by Type of Peginterferon and Genotype in Per Protocol Population Over Time
Description: Modified virological response (mVR) is defined as HCV RNA <50 IU/mL as assessed by CAP/CTM or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (LLOD 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The mVR is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment. PEOT= Post End of Treatment
Time Frame: At Week 2, Week 4, Week 12, EOT, and at 12 Weeks after EOT
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 564 | 231 | 151 | 16 | 3 | 2
percentage of participants
  Wk2, Peg IFN Alfa 2a (n=476,190,123,14,2,1) | 7.8 [5.5 to 10.6] | 32.1 [25.5 to 39.2] | 28.5 [20.7 to 37.3] | 21.4 [4.7 to 50.8] | 50.0 [1.3 to 98.7] | 100.0 [2.5 to 100.0]
  Wk2, Peg IFN Alfa 2b (n=88,41,28,2,1,1) | 3.4 [0.7 to 9.6] | 19.5 [8.8 to 34.9] | 32.1 [15.9 to 52.4] | 0.0 [0.0 to 84.2] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk4, Peg IFN Alfa 2a (n=476,190,123,14,2,1) | 25.4 [21.6 to 29.6] | 89.5 [84.2 to 93.5] | 83.7 [76.0 to 89.8] | 42.9 [17.7 to 71.1] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk4, Peg IFN Alfa 2b (n=88,41,28,2,1,1) | 23.9 [15.4 to 34.1] | 82.9 [67.9 to 92.8] | 75.0 [55.1 to 89.3] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk12, Peg IFN Alfa 2a (n=476,190,123,14,2,1) | 58.8 [54.3 to 63.3] | 98.4 [95.5 to 99.7] | 94.3 [88.6 to 97.7] | 71.4 [41.9 to 91.6] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk12,Peg IFN Alfa 2b (n=88,41,28,2,1,1) | 45.5 [34.8 to 56.4] | 95.1 [83.5 to 99.4] | 92.9 [76.5 to 99.1] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  EOT, Peg IFN Alfa 2a (n=476,190,123,14,2,1) | 56.5 [51.9 to 61.0] | 90.0 [84.8 to 93.9] | 81.3 [73.3 to 87.8] | 64.3 [35.1 to 87.2] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  EOT, Peg IFN Alfa 2b (n=88,41,28,2,1,1) | 44.3 [33.7 to 55.3] | 85.4 [70.8 to 94.4] | 71.4 [51.3 to 86.8] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  12wk PEOT,PegIFNAlfa2a(n=476,190,123,14,2,1) | 35.9 [31.6 to 40.4] | 63.2 [55.9 to 70.0] | 52.8 [43.6 to 61.9] | 42.9 [17.7 to 71.1] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  12wk PEOT, PegIFNAlfa2b(n=88,41,28,2,1,1) | 30.7 [21.3 to 41.4] | 51.2 [35.1 to 67.1] | 42.9 [24.5 to 62.8] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 97.5]

11. Secondary Outcome: Percentage of Participants With at Least a 2-log10 Drop in Hepatitis C Virus Ribonucleic Acid in Modified All Treated Population at Week 2, Week 4 and Week 12
Description: Participants with 2-logarithm (log) drop in HCV RNA including HCV RNA values <50 IU/mL in the serum from baseline to Week 2, Week 4 and Week 12, expressed in terms of a logarithmic scale with base 10 were evaluated and reported. A 2 log drop in HCV RNA was defined as drop of HCV viral load by 99%. The 2 log drop in HCV RNA is reported in treatment naive HCV mono-infected mTRT population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b.
Time Frame: At Week 2, Week 4 and Week 12
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 674 | 267 | 188 | 18 | 3 | 2
percentage of participants
  Wk2, Peg IFN Alfa 2a (n=568,221,159,16,2,1) | 19.9 [16.7 to 23.4] | 53.8 [47.0 to 60.6] | 48.4 [40.4 to 56.5] | 25.0 [7.3 to 52.4] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk2, Peg IFN Alfa 2b (n=106,46,29,2,1,1) | 17.0 [10.4 to 25.5] | 43.5 [28.9 to 58.9] | 62.1 [42.3 to 79.3] | 50.0 [1.3 to 98.7] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk4, Peg IFN Alfa 2a (n=568,221,159,16,2,1) | 53.7 [49.5 to 57.9] | 95.9 [92.4 to 98.1] | 92.5 [87.2 to 96.0] | 50.0 [24.7 to 75.3] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk4, Peg IFN Alfa 2b (n=106,46,29,2,1,1) | 43.4 [33.8 to 53.4] | 95.7 [85.2 to 99.5] | 86.2 [68.3 to 96.1] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk12, Peg IFN Alfa 2a (n=568,221,159,16,2,1) | 78.3 [74.7 to 81.7] | 99.5 [97.5 to 100.0] | 94.3 [89.5 to 97.4] | 62.5 [35.4 to 84.8] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk12,Peg IFN Alfa 2b (n=106,46,29,2,1,1) | 67.9 [58.2 to 76.7] | 97.8 [88.5 to 99.9] | 96.6 [82.2 to 99.9] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]

12. Secondary Outcome: Percentage of Participants With at Least a 2-log10 Drop in Hepatitis C Virus Ribonucleic Acid in Per Protocol Population at Week 2, Week 4 and Week 12
Description: Participants with 2-log drop in HCV RNA including HCV RNA values <50 IU/mL in the serum from baseline to Week 2, Week 4 and Week 12, expressed in terms of a logarithmic scale with base 10 were evaluated and reported. A 2 log drop in HCV RNA was defined as drop of HCV viral load by 99%. The 2 log drop in HCV RNA is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b.
Time Frame: At Week 2, Week 4 and Week 12
Population: Th PP population included all participants who met the inclusion and exclusion criteria of the study. n = the number of participants analyzed at a given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 564 | 231 | 151 | 16 | 3 | 2
percentage of participants
  Wk2, Peg IFN Alfa 2a (n=476,190,123,14,2,1) | 21.0 [17.4 to 24.9] | 57.4 [50.0 to 64.5] | 52.0 [42.8 to 61.1] | 28.6 [8.4 to 58.1] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk2, Peg IFN Alfa 2b (n=88,41,28,2,1,1) | 19.3 [11.7 to 29.1] | 46.3 [30.7 to 62.6] | 64.3 [44.1 to 81.4] | 50.0 [1.3 to 98.7] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk4, Peg IFN Alfa 2a (n=476,190,123,14,2,1) | 54.6 [50.0 to 59.2] | 98.4 [95.5 to 99.7] | 96.7 [91.9 to 99.1] | 57.1 [28.9 to 82.3] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk4, Peg IFN Alfa 2b (n=88,41,28,2,1,1) | 47.7 [37.0 to 58.6] | 95.1 [83.5 to 99.4] | 85.7 [67.3 to 96.0] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk12, Peg IFN Alfa 2a (n=476,190,123,14,2,1) | 79.6 [75.7 to 83.2] | 100.0 [98.1 to 100.0] | 98.4 [94.2 to 99.8] | 71.4 [41.9 to 91.6] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk12,Peg IFN Alfa 2b (n=88,41,28,2,1,1) | 72.7 [62.2 to 81.7] | 97.6 [87.1 to 99.9] | 96.4 [81.7 to 99.9] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]

13. Secondary Outcome: Percentage of Participants With at Least a 1-log10 Drop in Hepatitis C Virus Ribonucleic Acid in Modified All Treated Population at Week 2, Week 4 and Week 12
Description: Participants with 1-log drop in HCV RNA including HCV RNA values <50 IU/mL in the serum from baseline to Week 2, Week 4 and Week 12, expressed in terms of a logarithmic scale with base 10 were evaluated and reported. A 1- log drop in HCV RNA was defined as drop of HCV viral load by 90%. The 1- log drop in HCV RNA was reported in treatment naive HCV mono-infected mTRT population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b.
Time Frame: At Week 2, Week 4 and Week 12
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 674 | 267 | 188 | 18 | 3 | 2
percentage of participants
  Wk2, Peg IFN Alfa 2a (n=568,221,159,16,2,1) | 29.2 [25.5 to 33.2] | 56.1 [49.3 to 62.8] | 50.9 [42.9 to 58.9] | 31.3 [11.0 to 58.7] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk2, Peg IFN Alfa 2b (n=106,46,29,2,1,1) | 26.4 [18.3 to 35.9] | 45.7 [30.9 to 61.0] | 62.1 [42.3 to 79.3] | 50.0 [1.3 to 98.7] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk4, Peg IFN Alfa 2a (n=568,221,159,16,2,1) | 73.4 [69.6 to 77.0] | 97.3 [94.2 to 99.0] | 95.0 [90.3 to 97.8] | 68.8 [41.3 to 89.0] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk4, Peg IFN Alfa 2b (n=106,46,29,2,1,1) | 62.3 [52.3 to 71.5] | 95.7 [85.2 to 99.5] | 89.7 [72.6 to 97.8] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]

14. Secondary Outcome: Percentage of Participants With at Least a 1-log10 Drop in Hepatitis C Virus Ribonucleic Acid in Per-Protocol Population at Week 2, Week 4 and Week 12
Description: Participants with 1-log drop in HCV RNA including HCV RNA values <50 IU/mL in the serum from baseline to Week 2, Week 4 and Week 12, expressed in terms of a logarithmic scale with base 10 were evaluated and reported. A 1- log drop in HCV RNA was defined as drop of HCV viral load by 90%. The 1- log drop in HCV RNA was reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b.
Time Frame: At Week 2, Week 4 and Week 12
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 564 | 231 | 151 | 16 | 3 | 2
percentage of participants
  Wk2, Peg IFN Alfa 2a (n=476,190,123,14,2,1) | 31.1 [27.0 to 35.5] | 59.5 [52.1 to 66.5] | 53.7 [44.4 to 62.7] | 35.7 [12.8 to 64.9] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk2, Peg IFN Alfa 2b (n=88,41,28,2,1,1) | 29.5 [20.3 to 40.2] | 48.8 [32.9 to 64.9] | 64.3 [44.1 to 81.4] | 50.0 [1.3 to 98.7] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk4, Peg IFN Alfa 2a (n=476,190,123,14,2,1) | 74.6 [70.4 to 78.4] | 99.5 [97.1 to 100.0] | 98.4 [94.2 to 99.8] | 78.6 [49.2 to 95.3] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk4, Peg IFN Alfa 2b (n=88,41,28,2,1,1) | 65.9 [55.0 to 75.7] | 95.1 [83.5 to 99.4] | 89.3 [71.8 to 97.7] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]
  Wk12, Peg IFN Alfa 2a (n=476,190,123,14,2,1) | 91.6 [88.7 to 93.9] | 100.0 [98.1 to 100.0] | 99.2 [95.6 to 100.0] | 85.7 [57.2 to 98.2] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]
  Wk12,Peg IFN Alfa 2b (n=88,41,28,2,1,1) | 83.0 [73.4 to 90.1] | 97.6 [87.1 to 99.9] | 96.4 [81.7 to 99.9] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 97.5]

15. Secondary Outcome: Percentage of Participants With Predictive Values of Virological Response on Modified Sustained Virological Response After Treatment Initiation in Modified All Treated Population
Description: The probability that a participant who developed VR by Wk 2 achieved mSVR at 24 weeks after EOT was called the PPV of the VR by Wk 4 for mSVR. The probability that a participant who failed to develop VR by Wk 4 and 12 and also failed to achieve mSVR at 24 weeks after EOT was called the NPV of the VR by Wk 4 and 12 for mSVR. Predictive Values of VR was reported in treatment naive HCV mono-infected mTRT population participants who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 674 | 267 | 188 | 18 | 3 | 2
percentage of participants
  Wk2, Peg IFNAlfa2a,PPV (n=568,221,159,16,2,1) | 45.9 [29.5 to 63.1] | 63.2 [49.3 to 75.6] | 54.5 [36.4 to 71.9] | 0.0 [0.0 to 84.2] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | 0.0 [0.0 to 97.5]
  Wk2,Peg IFNAlfa2a,NPV (n=568,221,159,16,2,1) | 69.5 [63.5 to 75.1] | 43.1 [31.4 to 55.3] | 64.9 [51.1 to 77.1] | 66.7 [29.9 to 92.5] | 0.0 [0.0 to 84.2] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk2, Peg IFNAlfa 2b, PPV (n=106,46,29,2,1,1) | 100.0 [29.2 to 100.0] | 62.5 [24.5 to 91.5] | 57.1 [18.4 to 90.1] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | 0.0 [0.0 to 97.5] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk2, Peg IFNAlfa 2b, NPV (n=106,46,29,2,1,1) | 78.8 [65.3 to 88.9] | 50.0 [23.0 to 77.0] | 58.3 [27.7 to 84.8] | 100.0 [2.5 to 100.0] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.

16. Secondary Outcome: Percentage of Participants With Predictive Values of Virological Response on Modified Sustained Virological Response After Treatment Initiation in Per Protocol Population
Description: The probability that a participant who developed VR by Wk 2 and achieved mSVR at 24 weeks after EOT was called the PPV of the VR by Wk 4 for mSVR. The probability that a participant who failed to develop VR by Wk 2 and also failed to achieve mSVR at 24 weeks after EOT was called the NPV of the VR by Wk 2 for mSVR. Predictive values of VR is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 564 | 231 | 151 | 16 | 3 | 2
percentage of participants
  Wk2, Peg IFNAlfa2a, PPV (n=476,190,123,14,2,1) | 48.6 [31.4 to 66.0] | 61.8 [47.7 to 74.6] | 51.7 [32.5 to 70.6] | 0.0 [0.0 to 84.2] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | 0.0 [0.0 to 97.5]
  Wk2, PegIFNAlfa2a, NPV(n=476,190,123,14,2,1) | 67.0 [60.3 to 73.2] | 33.3 [21.7 to 46.7] | 56.1 [39.7 to 71.5] | 57.1 [18.4 to 90.1] | 0.0 [0.0 to 84.2] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk2, PegIFNAlfa2b, PPV(n=88,41,28,2,1,1) | 100.0 [29.2 to 100.0] | 62.5 [24.5 to 91.5] | 57.1 [18.4 to 90.1] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | 0.0 [0.0 to 97.5] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.
  Wk2, PegIFNAlfa2b, NPV(n=88,41,28,2,1,1) | 77.3 [62.2 to 88.5] | 53.8 [25.1 to 80.8] | 58.3 [27.7 to 84.8] | 100.0 [2.5 to 100.0] | NA [NA to NA] — Predictive values could not be determined as the denominator was zero. | NA [NA to NA] — Predictive values could not be determined as the denominator was zero.

17. Secondary Outcome: Number of Participants With Response by Disjoint Categories in Modified All-Treated Population at Week 4 and Week 12
Description: Rapid virological response (RVR) was defined as VR by Wk 4, Modified rapid virological response (mRVR) was defined as mVR by Wk 4, complete early virological response (cEVR) was defined as VR by Wk 12, but no RVR, modified complete early virological response (mcEVR) was defined as mVR by Wk 12, but no mRVR, partial early virological response (pEVR) was defined as at least a 2-log10 drop in HCV RNA as compared to baseline (including HCV RNA values <50 IU/mL) by Wk 12, but no RVR and no cEVR, modified partial early virological response (mpEVR) was defined as at least a 2-log10 drop in HCV RNA as compared to baseline by Wk 12, but no mRVR and no mcEVR. The data is reported in treatment naive HCV mono-infected mTRT participants who received PEG-IFN alfa-2a and PEG-IFN alfa-2b.
Time Frame: At Week 4 and Week 12
Population: The mTRT population included all participants who received at least one dose of PEG-IFN and ribavirin, and had at least one post-baseline HCV ribonucleic acid (RNA) result. Participants with a baseline result <50 IU/mL were excluded. n = the number of participants analyzed at a given time point.
Measure: Number; unit: participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 674 | 267 | 188 | 18 | 3 | 2
participants
  Peg IFN Alfa 2a RVR(n= 568,221,159,16,2,1) | 130 | 184 | 114 | 5 | 1 | 1
  Peg IFN Alfa 2b RVR (n= 106,46,29,2,1,1) | 19 | 38 | 20 | 2 | 1 | 0
  Peg IFN Alfa 2a mRVR(n= 568,221,159,16,2,1) | 147 | 189 | 120 | 6 | 2 | 1
  Peg IFN Alfa 2b mRVR(n= 106,46,29,2,1,1) | 24 | 39 | 22 | 2 | 1 | 0

18. Secondary Outcome: Number of Participants With Response by Disjoint Categories in Per-Protocol Population at Week 4 and Week 12
Description: RVR was defined as as VR by Wk 4, mRVR was defined as mVR by Wk 4, cEVR was defined as VR by Wk 12, but no RVR, mcEVR was defined as mVR by Wk 12, but no mRVR, pEVR was defined as at least a 2-log10 drop in HCV RNA as compared to baseline (including HCV RNA values <50 IU/mL) by Wk 12, but no RVR and no cEVR, mpEVR was defined as at least a 2-log10 drop in HCV RNA as compared to baseline by Wk 12, but no mRVR and no mcEVR. The data is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b.
Time Frame: During first 12 weeks of treatment
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 564 | 231 | 151 | 16 | 3 | 2
participants
  RVR, Peg IFN Alfa 2a (n=476,190,123,14,2,1) | 109 | 165 | 100 | 5 | 1 | 1
  RVR, Peg IFN Alfa 2b(n=88,41,28,2,1,1) | 16 | 33 | 19 | 2 | 1 | 0
  mRVR,Peg IFN Alfa 2a(n=476,190,123,14,2,1) | 121 | 170 | 103 | 6 | 2 | 1
  mRVR, Peg IFN Alfa 2b(n=88,41,28,2,1,1) | 21 | 34 | 21 | 2 | 1 | 0
  cEVR, Peg IFN Alfa 2a(n=476,190,123,14,2,1) | 155 | 21 | 15 | 5 | 1 | 0

19. Secondary Outcome: Percentage of Participants With Relapse After Modified End of Treatment Response by Genotype in Modified All-Treated Population at 12 Weeks After End of Treatment
Description: Participants whose last test result in their respective follow-up time window showed mVR were considered to have maintained their modified end of treatment response (mEOT-R). Participants whose last test result in the respective follow-up time window did not show mVR, or who did not have a test result in the respective follow-up time window but whose last follow-up test result before the time window did not show mVR, were considered to have relapsed. Only participants with mEOT-R who had a HCV RNA measurement in the follow-up time window (without use of backward imputation), or whose last HCV RNA measurement at a follow-up time point before the time window did not show mVR, were included in the calculations. The number of participants with relapse was reported in treatment naive mTRT population who received PEG-IFN alfa-2a and PEG-IFN alfa-2b. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 12 weeks after EOT
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 172 | 112 | 72 | 6 | 1 | 1
Percentage of Participants
  12wk PEOT,PegIFN Alfa2a (n=153,94,63,4,1,1) | 24.8 | 8.5 | 22.2 | 0.0 | 0.0 | 0.0
  12wk PEOT, PegIFN Alfa2b(n=19,18,9,2,0,0) | 10.5 | 11.1 | 0.0 | 0.0 | NA — There were no participants with an mVR who also had a HCV RNA test at the 12 weeks after EOT follow-up time point for G5/6 and UNK genotype subgroups. | NA — There were no participants with an mVR who also had a HCV RNA test at the 12 weeks after EOT follow-up time point for G5/6 and UNK genotype subgroups.

20. Secondary Outcome: Percentage of Participants With Relapse After Modified End of Treatment Response by Genotype in Modified All-Treated Population at 24 Weeks After End of Treatment
Description: Participants whose last test result in the follow-up time window showed mVR were considered to have maintained their modified end of treatment response (mEOT-R). Participants whose last test result in the respective follow-up time window did not show mVR, or who did not have a test result in the respective follow-up time window but whose last follow-up test result before the time window did not show mVR, were considered to have relapsed. Only participants with mEOT-R who had a HCV RNA measurement in the follow-up time window (without use of backward imputation), or whose last HCV RNA measurement at a follow-up time point before the time window did not show mVR, were included in the calculations. It was reported in treatment naive HCV mono-infected mTRT population receiving PEG-IFN alfa-2a and PEG-IFN alfa-2b. EOT= 12, 24, 48 or 72 weeks after initiation of treatment. No participants were analysed for arm 'Genotype Unknown'.
Time Frame: 24 weeks after EOT
Population: as for outcome 17
Measure: Number; unit: Percentage of Participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 264 | 161 | 95 | 7 | 3 | 0
Percentage of Participants
  24wk PEOT,PegIFN Alfa2a (n=236,136,84, 6, 2, 0) | 26.3 | 8.8 | 19.0 | 16.7 | 0.0 |
  24wk PEOT, PegIFN Alfa2b(n=28, 25, 11, 1, 1, 0) | 10.7 | 8.0 | 0.0 | 0.0 | 100.0 |
Statistical Analysis 1: Comparison: Genotype 1 (G1); The statistical analysis is presented for Sex (MALE vs FEMALE). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0162, Regression, Logistic; Odds Ratio (OR) = 0.441, 95% CI 2-sided [0.226 to 0.859]
Statistical Analysis 2: Comparison: Genotype 1 (G1); The statistical analysis is presented for HCV RNA at BL in log10(IU/mL). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0156, Regression, Logistic; Odds Ratio (OR) = 1.745, 95% CI 2-sided [1.111 to 2.741]
Statistical Analysis 3: Comparison: Genotype 1 (G1); The statistical analysis is presented for Alanine Aminotransferase (ALT) ratio at BL (<=1 vs > 3). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.1075, Regression, Logistic; Odds Ratio (OR) = 2.372, 95% CI 2-sided [0.829 to 6.789]
Statistical Analysis 4: Comparison: Genotype 1 (G1); The statistical analysis is presented for ALT ratio at BL (> 1 - 3 vs > 3). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.8518, Regression, Logistic; Odds Ratio (OR) = 0.906, 95% CI 2-sided [0.321 to 2.559]
Statistical Analysis 5: Comparison: Genotype 1 (G1); The statistical analysis is presented for treatment duration after VR in weeks. The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Wk 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0012, Regression, Logistic; Odds Ratio (OR) = 0.969, 95% CI 2-sided [0.951 to 0.988]
Statistical Analysis 6: Comparison: Genotype 1 (G1); The statistical analysis is presented for Sex (MALE vs FEMALE). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0162, Regression, Logistic; Odds Ratio (OR) = 0.441, 95% CI 2-sided [0.226 to 0.859]
Statistical Analysis 7: Comparison: Genotype 1 (G1); The statistical analysis is presented for HCV RNA at BL in log10(IU/mL). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0156, Regression, Logistic; Odds Ratio (OR) = 1.745, 95% CI 2-sided [1.111 to 2.741]
Statistical Analysis 8: Comparison: Genotype 1 (G1); The statistical analysis is presented for ALT ratio at BL (<=1 vs > 3). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.1075, Regression, Logistic; Odds Ratio (OR) = 2.372, 95% CI 2-sided [0.829 to 6.789]
Statistical Analysis 9: Comparison: Genotype 1 (G1); The statistical analysis is presented for ALT ratio at BL (> 1 - 3 vs > 3). The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.8518, Regression, Logistic; Odds Ratio (OR) = 0.906, 95% CI 2-sided [0.321 to 2.559]
Statistical Analysis 10: Comparison: Genotype 1 (G1); The statistical analysis is presented for treatment duration after VR in weeks. The logistic regression analysis for relapse was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0012, Regression, Logistic; Odds Ratio (OR) = 0.969, 95% CI 2-sided [0.951 to 0.988]
Statistical Analysis 11: Comparison: Genotype 2 (G2); [analysis description as in outcome 20, analysis 5]; Test type: Superiority or Other; p = 0.0017, Regression, Logistic; Odds Ratio (OR) = 0.848, 95% CI 2-sided [0.765 to 0.940]
Statistical Analysis 12: Comparison: Genotype 2 (G2); [analysis description as in outcome 20, analysis 10]; Test type: Superiority or Other; p = 0.0017, Regression, Logistic; Odds Ratio (OR) = 0.848, 95% CI 2-sided [0.765 to 0.940]
Statistical Analysis 13: Comparison: Genotype 1 (G1); The statistical analysis is presented for Sex (MALE vs FEMALE). The logistic regression analysis for relapse was performed for association between treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0071, Regression, Logistic; Odds Ratio (OR) = 0.401, 95% CI 2-sided [0.206 to 0.780]
Statistical Analysis 14: Comparison: Genotype 1 (G1); The statistical analysis is presented for On-treatment response (RVR vs NO RVR/EVR). The logistic regression analysis for relapse was performed for association between treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 0.016, 95% CI 2-sided [0.001 to 0.169]
Statistical Analysis 15: Comparison: Genotype 1 (G1); The statistical analysis is presented for On-treatment response (cEVR vs NO RVR/EVR). The logistic regression analysis for relapse was performed for association between treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0255, Regression, Logistic; Odds Ratio (OR) = 0.076, 95% CI 2-sided [0.008 to 0.729]
Statistical Analysis 16: Comparison: Genotype 1 (G1); The statistical analysis is presented for On-treatment response (pEVR vs NO RVR/EVR). The logistic regression analysis for relapse was performed for association between treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.1501, Regression, Logistic; Odds Ratio (OR) = 0.184, 95% CI 2-sided [0.018 to 1.845]
Statistical Analysis 17: Comparison: Genotype 2 (G2); The statistical analysis is presented for On-treatment response (cEVR vs RVR). The logistic regression analysis for relapse was performed for association between treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 27.250, 95% CI 2-sided [6.729 to 110.35]

21. Secondary Outcome: Percentage of Participants With Relapse After Modified End of Treatment Response by Genotype in Per-Protocol Population at 12 Weeks After End of Treatment
Description: Participants whose last test result in the follow-up time window showed mVR were considered to have maintained their modified end of treatment response (mEOT-R). Participants whose last test result in the respective follow-up time window did not show mVR, or who did not have a test result in the respective follow-up time window but whose last follow-up test result before the time window did not show mVR, were considered to have relapsed. Only participants with mEOT-R who had a HCV RNA measurement in the follow-up time window (without use of backward imputation), or whose last HCV RNA measurement at a follow-up time point before the time window did not show mVR, were included in the calculations. It was reported in treatment naive HCV mono-infected PP population receiving PEG-IFN alfa-2a and PEG-IFN alfa-2b. EOT= 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 12 weeks after EOT
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 144 | 101 | 63 | 6 | 1 | 1
Percentage of Participants
  12wk PEOT,PegINFAlfa2a (n=128,86,55,4,1,1) | 23.4 | 8.1 | 21.8 | 0.0 | 0.0 | 0.0
  12wk PEOT, PegIFNAlfa2b(n=16,15,8,2,0,0) | 12.5 | 13.3 | 0.0 | 0.0 | NA — There were no participants with an mVR who also had a HCV RNA test at the 12 weeks after EOT follow-up time point for G5/6 and UNK genotype subgroups. | NA — There were no participants with an mVR who also had a HCV RNA test at the 12 weeks after EOT follow-up time point for G5/6 and UNK genotype subgroups.

22. Secondary Outcome: Percentage of Participants With Relapse After Modified End of Treatment Response by Genotype in Per-Protocol Population at 24 Weeks After End of Treatment
Description: Participants whose last test result in the follow-up time window showed mVR were considered to have maintained their modified end of treatment response (mEOT-R). Participants whose last test result in the respective follow-up time window did not show mVR, or who did not have a test result in the respective follow-up time window but whose last follow-up test result before the time window did not show mVR, were considered to have relapsed. Only participants with mEOT-R who had a HCV RNA measurement in the follow-up time window (without use of backward imputation), or whose last HCV RNA measurement at a follow-up time point before the time window did not show mVR, were included in the calculations. It was reported in treatment naive HCV mono-infected PP population receiving PEG-IFN alfa-2a and PEG-IFN alfa-2b. EOT= 12, 24, 48 or 72 weeks after initiation of treatment. No participants were analysed for arm 'Genotype Unknown'.
Time Frame: At 24 weeks after EOT
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Genotype 1 (G1) | Genotype 2 (G2) | Genotype 3 (G3) | Genotype 4 (G4) | Genotype 5/6 (G5/6) | Genotype Unknown (UNK)
Number analyzed (Participants) | 227 | 142 | 82 | 7 | 3 | 0
Percentage of Participants
  24wk PEOT,PegIFNAlfa2a (n=201, 120, 72, 6, 2, 0) | 24.4 | 8.3 | 18.1 | 16.7 | 0.0 |
  24wk PEOT, PegIFNAlfa2b(n=26,22,10,1,1, 0) | 11.5 | 9.1 | 0.0 | 0.0 | 100.0 |

ADVERSE EVENTS:
Time Frame: Up to 3 years and 8 months
Description: An Adverse events (AE) was any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. The safety population included all participants who received at least one dose of either PEG-IFN or ribavirin.
Groups:
- Total (PEG-IFN Alfa-2a +PEG-IFN Alfa-2b): Eligible participants with serologically proven CHC who received PEG-IFN alfa-2a or PEG-IFN alfa-2b plus ribavirin for up to 48 weeks according to the standard of care and in line with SPCs/local labeling were observed.
Arm/Group | Total (PEG-IFN Alfa-2a +PEG-IFN Alfa-2b)
Serious Adverse Events (participants affected / at risk) | 130/1441
Other Adverse Events (participants affected / at risk) | 841/1441
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total (PEG-IFN Alfa-2a +PEG-IFN Alfa-2b) (N=1441)
Pneumonia (Infections and infestations) | 10
Cellulitis (Infections and infestations) | 3
Appendicitis (Infections and infestations) | 1
Appendicitis perforated (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Peritonitis bacterial (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Salmonellosis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sepsis syndrome (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Depression (Psychiatric disorders) | 5
Alcoholism (Psychiatric disorders) | 3
Psychotic disorder (Psychiatric disorders) | 3
Suicidal ideation (Psychiatric disorders) | 3
Suicide attempt (Psychiatric disorders) | 3
Mental status changes (Psychiatric disorders) | 2
Acute psychosis (Psychiatric disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression suicidal (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 10
Pancytopenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Bicytopenia (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Abdominal adhesions (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Overdose (Injury, poisoning and procedural complications) | 3
Ankle fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Gun shot wound (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Chest pain (General disorders) | 5
Chest discomfort (General disorders) | 1
Death (General disorders) | 1
Fatigue (General disorders) | 1
Impaired healing (General disorders) | 1
Irritability (General disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3
Diabetes mellitus inadequate Control (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 4
Convulsion (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Toxic encephalopathy (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
Phlebitis superficial (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal failure acute (Renal and urinary disorders) | 3
Nephrolithiasis (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Chronic hepatic failure (Hepatobiliary disorders) | 1
Hepatic lesion (Hepatobiliary disorders) | 1
Blood glucose increased (Investigations) | 1
Laboratory test interference (Investigations) | 1
Platelet count decreased (Investigations) | 1
Cataract (Eye disorders) | 1
Scleritis (Eye disorders) | 1
Drug rehabilitation (Surgical and medical procedures) | 1
Hysterectomy (Surgical and medical procedures) | 1
Fanconi Syndrome (Congenital, familial and genetic disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Ovarian mass (Reproductive system and breast disorders) | 1
Substance use (Social circumstances) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total (PEG-IFN Alfa-2a +PEG-IFN Alfa-2b) (N=1441)
Depression (Psychiatric disorders) | 234
Insomnia (Psychiatric disorders) | 224
Anxiety (Psychiatric disorders) | 92
Anaemia (Blood and lymphatic system disorders) | 333
Neutropenia (Blood and lymphatic system disorders) | 108
Fatigue (General disorders) | 206
Influenza like illness (General disorders) | 104
Irritability (General disorders) | 74
Rash (Skin and subcutaneous tissue disorders) | 138
Pruritus (Skin and subcutaneous tissue disorders) | 80
Nausea (Gastrointestinal disorders) | 168
Myalgia (Musculoskeletal and connective tissue disorders) | 78
Arthralgia (Musculoskeletal and connective tissue disorders) | 75
Headache (Nervous system disorders) | 136
Decreased appetite (Metabolism and nutrition disorders) | 79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.